CLINICAL TRIAL: NCT04554537
Title: Strategic Memory and Reasoning Training for Cognitive Problems Due to Mild Traumatic Brain Injury and Posttraumatic Stress Disorder
Brief Title: Strategic Memory and Reasoning Training for Cognitive Problems
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Kristin Samuelson (Other)
Responsible Party: Sponsor-Investigator, Dr. Kristin Samuelson, Associate Professor of Psychology, University of Colorado, Colorado Springs
Organization: University of Colorado, Colorado Springs (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMART
Record Dates: First submitted 2020-01-09; First posted 2020-09-18 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Traumatic Brain Injury; Posttraumatic Stress Disorder
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain Health Workshop (Placebo Comparator): The BHW training has been used in multiple prior studies as a comparison training program in cognitive training trials It consists of sessions of fact-based information about the brain but does not train cognitive strategies. Topics include neuroanatomy, neuroplasticity, and effects of TBI on cognitive functioning. Other sessions focus on diet, exercise, sleep, and social functioning and their relationships to brain health. Participants are encouraged to share how the topics impact their lives. Participants are given take-home reading materials on related topics that were then discussed at the last session. At home, they were instructed to watch assigned videos but had no other homework.
  Interventions: Behavioral: Brain Health Workshop
- SMART (Experimental): SMART emphasizes top-down processing by targeting focused attention, assimilation of information, and mental flexibility and innovation, all higher-order cognitive functions driven by the frontal lobes. SMART was delivered in small groups (n = 2 to 8) consisting of two 3-hour sessions over two days, followed by one 3-hour session a month later. Overall, sessions focused on strategic attention, integrative reasoning, and cognitive control functions (Chapman, 2014). Training consists of initial sessions of skills training with the one-month follow-up session being a "booster session" consisting of review. We modified the training such that all sessions included skills training with briefer review. The first two sessions consisted of strategic attention and integrated reasoning and the final session discussed innovation.
  Interventions: Behavioral: SMART

INTERVENTIONS:
Behavioral: SMART — A treatment program developed to address specific brain functions found to be crucial for the recovery following brain injury.
  Other Names: Strategic Memory Advanced Reasoning Training
  Arms: SMART
Behavioral: Brain Health Workshop — A psychoeducation program designed to provide in depth information to participants about the neuroscience behind their TBI and PTSD and the symptoms and challenges they may experience.
  Arms: Brain Health Workshop

SUMMARY:
The focus of this study is to test a treatment program (Strategic Memory Advanced Reasoning Training; SMART) that was developed to address specific brain functions found to be crucial for the recovery following traumatic brain injury (TBI). New research has shown that when these very specific brain functions are targeted, such as ability to focus on a task while ignoring irrelevant information, brain changes are more significant. SMART emphasizes top-down processing by targeting focused attention, assimilation of information, and mental flexibility and innovation, all higher-order cognitive functions driven by the frontal lobes. Evidence from other top-down cognitive training programs demonstrates their effectiveness in improving cognitive and daily functioning in individuals reporting a TBI. In addition to improving frontal lobe capacity, SMART has also been shown to increase brain blood flow critical for complex thinking and strengthen white matter integrity. The effectiveness of SMART has been extensively tested with a variety of populations, including healthy adults and adolescents, adolescents with brain injuries, healthy seniors and those at risk for Alzheimers, and veterans and civilians with lingering impairment following TBIs. This will be the first study to test its effectiveness with individuals with mild TBI (MTBI) and posttraumatic stress disorder (PTSD).

The SMART program has previously been tested with patients with TBI using an 18-hour training format. When compared to the Brain Health Workshop (BHW), an education-based active learning module, participants in the SMART group (n = 31) demonstrated improvements in gist reasoning, executive function, and memory, generalization of improvement to daily functioning activities and continuation of these gains 6 months posttraining. The training consisted of 15 hours of training conducted over 10 group sessions in the first 5 weeks and a final 3 hours of training at spaced intervals over the next 3 weeks. SMART training has not been tested with patients with PTSD-related neuropsychological impairments. The purpose of the current study is to investigate the efficacy of a shortened training program (9 hours) in improving neurocognitive function in patients with mTBI and/or PTSD.

DETAILED DESCRIPTION:
DESIGN: This is a double-blind, randomized controlled clinical trial. A total of 150 adults ages 19-65 years with Traumatic Brain Injury (TBI) and/or subthreshold of full diagnosis of posttraumatic stress disorder (PTSD) will be recruited for the study (estimated 100 completers). They will be read the telephone recruitment script (attached) and asked questions that determine whether or not they are eligible for the study. Eligible participants will be randomized into either SMART training or the Brain Health Workshop as a control condition. All the participants will go through the neuropsychological testing and clinical interviews before and after the treatment program and six months later to assess long terms changes. These testing procedures are explained below. During the treatment program, SMART participants will participate in a 6-hour program over a 1-week period (two 3-hour sessions), and one 3-hour booster session a month later. Participants in the Brain Health Workshop condition will attend sessions that include education on brain topics of the same duration. TESTING SESSIONS: Participants will attend an initial eligibility visit and a second visit in which they will complete neuropsychological tests. They will also complete a packet of self-report questionnaires at home in between the first two visits (listed in section 2c below). At the initial eligibility visit, they will met with a clinical interviewer/neuropsychological technician (a graduate student working under Dr. Samuelson's supervision) who will administer the following measures:Clinician-Administered PTSD Scale (CAPS),Brief Pain Inventory - Short Form (BPI-SF), Glasgow Outcome Scale - Extended (GOSE),Ohio State University TBI Identification Method (OSU-TBI-ID), NIH Toolbox Standing Balance Test (motor),and Test of Memory Malingering Trial. These measures will determine eligibility for the study (i.e., diagnosis of TBI and/or subthreshold or full PTSD, no diagnosis of psychosis, bipolar disorder, or substance dependence, and no malingering). At the second visit, the technician will administer neuropsychological tests , which will take 2.5 to 3 hours: Wechsler Adult Intelligence Scale-IV (WAIS-IV) Coding, WAIS-IV Symbol Search, WAIS-IV Digit Span, Wechsler Memory Scale-IV (WMS-IV) Logical Memory, Test of Strategic Learning (TOSL),Visual Selective Learning Task, Go/No-Go, WMS-IV Logical Memory II, WAIS-IV Vocabulary, WAIS-IV Similarities, WAIS-IV Matrix Reasoning, Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency Test, D-KEFS Color-Word Interference Test , D-KEFS Trail Making Test, Brief Visuospatial Memory Test - Revised (BVMT), Rey Complex Figure Test & Recognition Trial (RCFT), Animal Fluency-Verbal, California Verbal Learning Test, Controlled Oral Word Association (COWAT) , Wide Range Achievement Test-4 (WRAT-4) Word Reading, Paced Auditory Serial Addition Test (PASAT). TREATMENT: Following baseline testing sessions, the participants will be randomly assigned to either SMART or Brain Health Workshop (BHW). In the SMART treatment condition, participants will be taught new strategies in a group setting to improve brain functions such as critical thinking, reasoning, problem solving and improved comprehension of information. To accomplish improvement in these brain functions, participants will be involved in activities such as analyzing information from a book, or a newspaper article, writing comprehensive passages etc. Training will also include application of these strategies to other daily activities. In this treatment group, participants will also be given homework assignments for each session including maintaining a journal, provided by the clinician to record the use of the strategies taught in the treatment sessions in their daily activities and the homework provided by the clinician. The intervention will be a total of 9 hours - 6 hours over the course of one week and then a 3-hour booster session a month later. Post-testing occurs within one week of the booster session. In the BHW condition, participants will be taught topics about the brain in a similar format to SMART. Topics include anatomy, neurotransmitters, effects of TBI on cognitive functioning, and principles of neuroplasticity. Participants will also be given take-home reading assignments and quizzed on the readings at the beginning of the following session. Post-Treatment: Following the interventions patients will repeat the assessments (except for Test of Memory Malingering (TOMM), and TBI interviews) identical to the pre-treatment assessment within one week of completing the intervention. This testing session will occur in 1 day and take approximately 3.25 to 4 hours. Participants will be tested again at 6 months following the intervention with the same tests.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria include .

* adults between the ages of 19 to 65 years
* speak and comprehend English, as not all of the standardized cognitive tests have been normed for non-English speakers
* diagnosis of either mild or moderate TBI (as defined by OSU TBI interview) and/or diagnosis of subthreshold or full PTSD (as determined by Clinician-Administered PTSD Scale)

Exclusion Criteria:

* someone who is not proficient in reading, comprehending, and speaking English
* self-report on phone screen interview of pre-existing cerebral palsy, intellectual disability, autism, epilepsy, schizophrenia, stroke, pervasive developmental disorder, or a diagnosed learning disability
* history of psychotic disorder or bipolar disorder (by self-report)
* current alcohol or drug dependence (by self-report)
* severe TBI (determined by OSU TBI interview)
* participants who are determined by the TOMM (more than five errors on Trial 2 or the Retention trial) to be malingering neuropsychological problems
* neuropsychological testing or r any cognitive training in the past 3 months as this could introduce practice effects.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
CHANGE in Digit Span test of the Wechsler Adult Intelligence Scale - Fourth Edition | Pre-training, immediately post-training and six months later
  Digit Span requires participants to repeat digits forwards, backwards, and sequences in ascending order; the combined score of these three tasks was used, which is then converted to a scaled score with a range of 1 to 19. Higher scores represent better performance.
CHANGE in Digit Symbol and Symbol Search tests, which comprise the Processing Speed Index of the WAIS-IV | Pre-training, immediately post-training and six months later
  To assess processing speed and visual-motor coordination. The Processing Speed Index is a standard score with a range of 50 to 150 with higher scores indicating better performance.
CHANGE in California Verbal Learning Test | Pre-training, immediately post-training and six months later
  Participants hear a word list over five trials and repeat back as many words as they can remember; the sum of trials 1-5 serves as a measure of immediate verbal memory and the delayed memory for the words 20 minutes later serves as a measure of delayed verbal memory. Scores are converted from raw scores to T scores. T scores have a range of 20 to 80, with higher scores representing bettery performance.
CHANGE in Logical Memory task of the Wechsler Memory Scale, 4th edition | Pre-training, immediately post-training and six months later
  assess verbal learning and memory in a narrative context. Participants were presented with a short story and asked to repeat back as much of the story as possible immediately after. Details of the stories are totaled and raw scores are converted to scaled scores. Both immediate memory and delayed memory received a scaled score, range from 1 to 19 with higher scores indicating better performance.
CHANGE in Brief Visuospatial Memory Test-Revised | Pre-training, immediately post-training and six months later
  a measure of immediate and delayed visuospatial memory. The participant must memorize a series of designs over three trials and recreate them from memory, both immediately following display and after a delay of 20 minutes. A sum of Trials 1-3 represents the immediate raw score which is then converted to a T score. The T scores have a range of 20 to 80, with higher scores indicating better performance.
CHANGE in Trail Making Test of the Delis-Kaplan Executive Functioning System | Pre-training, immediately post-training and six months later
  Assess cognitive flexibility, verbal fluency, inhibitory control. There are five conditions, and the final condition, the "switching condition" is the score used. It is a measure of seconds taken to complete the task which is then converted to a scaled score, with a range of 1 to 19, with higher scores representing better performance.
CHANGE in Test of Strategic Learning | Pre-training, immediately post-training and six months later
  The TOSL involves synthesizing gist meaning from complex information. Participants read a complex passage and are instructed to generate a high-level summary of what they read. Three scores are generated and are presented as raw scores, with higher scores indicating better performance. The summary abstraction score reflects the total number of accurately abstracted meanings from the reading; the high-level lessons score measures the number of high-level lessons the participants gleaned from the story; and the detail total score measures participants' memory for the story's detail-based information.
CHANGE in Neurobehavioral Symptom Inventory (NSI) | Pre-training, immediately post-training and six months later
  22-item self-report measure of postconcussive symptoms. We specifically examined the Cognitive subscale of the NSI at all time points. The range for this scale is 0 to 20, with higher scores indicating more self-reported impairment
CHANGE in Clinician Administered PTSD Scale for Diagnostic and Statistical Manual (DSM)-5 | Pre-training, immediately post-training and six months later
  Assesses posttraumatic stress diagnosis and symptoms. Range of scores is 0 to 80 with higher scores indicating higher PTSD symptom severity.
CHANGE in Paced Auditory Serial Addition Test | Pre-training, immediately post-training and six months later
  To assess working memory, sustained attention, and divided attention, participants were asked to listen to an audio tape presenting a series of single-digit numbers and then state aloud the sum of the number more recently presented plus the number preceding it. There were two trials and the number of correct answers for both trials is summed. Higher scores indicated better performance.
CHANGE in Continuous Performance Test performance | Pre-training, immediately post-training and six months later
  To assess sustained attention, vigilance, inhibitory control, and inattention, the computer-based Conners' Continuous Performance Test 3rd Edition was administered. Errors of omission are a measure of sustained attention and errors of commission are a measure of inhibitory control. Raw scores are converted to T scores. Higher scores indicate more omissions and commissions, or poorer performance.
CHANGE in Delis-Kaplan Executive Functioning System Color-Word Interference Test performance | Pre-training, immediately post-training and six months later
  To assess change in inhibitory control and cognitive flexibility, the "interference condition" of the Color-Word Test was used. Raw scores are converted to scaled scores, with a range of 1 to 19 with higher scores representing better performance.
CHANGE in Delis-Kaplan Executive Functioning System Verbal Fluency performance | Pre-training, immediately post-training and six months later
  To assess change in verbal fluency, two tasks were administered: the Letter Fluency subtest and the Category Fluency subtest. Raw scores are converted into scaled scores, with a range of 1 to 19 with higher scores representing better performance.

SECONDARY OUTCOMES:
Change in subjective cognitive complaints | Pre-training, immediately post-training and six months later
  To assess change in subjective cognitive complaints, the Cognitive Self-Report Questionnaire was administered. Total score from the cognitive subscale will be used, with scores ranging from 12 to 60. Higher scores represent more cognitive complaints.
Change in Quality of Life | Pre-training, immediately post-training and six months later
  To assess change in quality of life, the World Health Organization Quality of Life Scale was administered. The total score was used, which ranges from 25 to 125, with higher scores indicating higher quality of life and functioning across domains

CONTACTS AND LOCATIONS:
Overall Officials: Kristin W Samuelson, PhD, Principal Investigator — UCCS

IPD SHARING:
Plan to Share IPD: No
There is not currently a plan to share individual participant data (IPD).